CLINICAL TRIAL: NCT01348919
Title: An Open-Label Study to Determine the Maximum Tolerated Dose and Evaluate the Safety and Efficacy of CEP-18770 in Combination With Lenalidomide and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Delanzomib (CEP-18770) in Combination With Lenalidomide and Dexamethasone in Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C18770/2049; 2010-020910-27 (EudraCT Number)
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-05

CONDITIONS: Multiple Myeloma
Keywords: Cancer; Multiple myeloma; CEP-18770; Lenalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — delanzomib; Lenalidomide; Dexamethasone

ARMS (3):
- CEP-18770 Dose A (Experimental): Participants will receive CEP-18770 Dose A intravenously (IV) on Days 1, 8, and 15 in each 28-day cycle. In addition, participants will receive a fixed dose of 25 mg oral lenalidomide on Days 1 through 21 and a fixed dose of 40 mg oral dexamethasone on Days 1, 8, 15, and 22 of each 28-day cycle.
  Interventions: Drug: CEP-18770; Drug: Lenalidomide; Drug: Dexamethasone
- CEP-18770 Dose B (Experimental): Participants will receive CEP-18770 Dose B IV on Days 1, 8, and 15 in each 28-day cycle. In addition, participants will receive a fixed dose of 25 mg oral lenalidomide on Days 1 through 21 and a fixed dose of 40 mg oral dexamethasone on Days 1, 8, 15, and 22 of each 28-day cycle.
  Interventions: Drug: CEP-18770; Drug: Lenalidomide; Drug: Dexamethasone
- CEP-18770 Dose C (Experimental): Participants will receive CEP-18770 Dose C IV on Days 1, 8, and 15 in each 28-day cycle. In addition, participants will receive a fixed dose of 25 mg oral lenalidomide on Days 1 through 21 and a fixed dose of 40 mg oral dexamethasone on Days 1, 8, 15, and 22 of each 28-day cycle.
  Interventions: Drug: CEP-18770; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: CEP-18770 — CEP-18770 will be administered per dose and schedule specified in the arm description.
  Other Names: Delanzomib
Drug: Lenalidomide — Lenalidomide will be administered per dose and schedule specified in the arm description.
Drug: Dexamethasone — Dexamethasone will be administered per dose and schedule specified in the arm description.

SUMMARY:
The primary objective of the study is to determine the maximum tolerated dose (MTD) of CEP-18770 in combination with lenalidomide and dexamethasone in participants with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
After cycle 1, the start of treatment in each cycle may occur within a 3-day window. In addition, after cycle 2, the start of treatment in cycle 3 may be delayed by 1 week if, in the opinion of the investigator, the delay is warranted. If a participant cannot receive 75% of the planned dose for any of the 3 agents (missing more than 1 dose of CEP-18770, or more than 5 doses of lenalidomide [either consecutively or separately], or more than 1 dose of dexamethasone [either consecutively or separately]), due to a drug-related adverse event, the event will be considered a dose limiting toxicity (DLT), even if the grade of toxicity is lower than specified DLT determination. Participants will receive intravenous (IV) CEP-18770 on Days 1, 8, and 15, oral lenalidomide on days 1 through 21, and oral dexamethasone on days 1, 8, 15, and 22 of each 28-day cycle. Treatment with all 3 drugs will continue for up to 12 cycles (approximately 11 months), or until disease progression or intolerable toxicities. Participants experiencing clinical benefit may continue to receive additional treatment at the investigator's discretion and following sponsor notification. In part 2 of the study, participants will receive CEP-18770 as a slow IV bolus (approximately 1 milliliter per minute) at the maximum tolerated dose on days 1, 8, and 15 of every 28-day cycle. Participants who complete or discontinue study drug treatment and whose disease has not progressed will have study visits every 7-9 weeks during follow-up until disease progression, death, or until they have been monitored for 1 year after the first administration of study drug, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* The participant is a man or woman at least 18 years of age with documented multiple myeloma.
* The participant has relapsed or progressive disease after receiving at least 1 previous chemotherapy treatment but no more than 5 previous therapies.
* The participant has measurable disease defined as 1 of the following:
* serum M-protein 0.5 grams (g)/deciliter (dL) or greater
* urine M-protein 200 mg/24 hours or greater
* The participant has a life expectancy of more than 3 months.
* Written informed consent is obtained.
* The participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* The participant has adequate hepatic and renal function and hematologic assessments as specified by the study protocol
* The participant has been independent of support with granulocyte-colony stimulating factor (G-CSF) or granulocyte macrophage-colony stimulating factor (GM-CSF) for more than 1 week at the time of screening.
* The participant has been independent of platelet transfusions for 1 week at the time of screening.
* The participant may have received an allogeneic and/or autologous transplant.
* The participant must agree to register into the mandatory risk evaluation and mitigation program for receiving lenalidomide if required by local regulations.
* Agreement by women of childbearing potential (not surgically sterile or 24 months postmenopausal) to use 2 medically accepted methods of contraception and must agree to continue use of these methods from 4 weeks prior to treatment to 4 weeks after treatment. Acceptable methods of contraception include at least one highly effective method (for example, intrauterine device [IUD], non-combination hormonal contraception, tubal ligation, or partner's vasectomy) and one additional method (for example, latex condom, diaphragm, or cervical cap).
* Agreement by men who are sexually active with a woman of childbearing potential (as defined in the criterion above), to use a condom during any sexual contact for the duration of the study and for 4 weeks after the last administration of study drug. This requirement applies even if the man has had a vasectomy.
* The participant may not donate blood, semen or sperm while taking lenalidomide or for 4 weeks after the last administration of lenalidomide.
* The participant may not breastfeed while taking lenalidomide or for 4 weeks after the last administration of lenalidomide.

Exclusion Criteria:

* The participant has nonmeasurable multiple myeloma, defined as less than 0.5 g/dL M-protein in the serum, and less than 200 mg/24 hours M-protein in the urine.
* The participant could not tolerate previous lenalidomide or low-dose dexamethasone treatment.
* The participant had previous treatment with CEP-18770.
* The participant has POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy or monoclonal proliferative disorder, and skin changes [increased skin pigment, increased body hair, thickening of the skin, whitening of the nails, etc]).
* The participant has plasma cell leukemia or primary amyloidosis.
* The participant received chemotherapy with approved or investigative anticancer therapeutics within 3 weeks before the first dose of study drug.
* The participant received radiation therapy or immunotherapy within 4 weeks or localized radiation therapy within 1 week prior to the first dose of study drug.
* The participant had major surgery within 3 weeks before the first dose of study drug.
* The participant has congestive heart failure (New York Heart Association Class III to IV) or had symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within the last 6 months.
* The participant had an acute infection requiring systemic antibiotics, antiviral agents, or antifungal agents within 2 weeks before the first dose of study drug.
* The participant has a known or suspected human immunodeficiency virus (HIV) infection, acute or chronic hepatitis B virus or hepatitis C virus on the basis of their medical history.
* The participant has myelodysplastic or myeloproliferative syndrome.
* The participant has significant neuropathy (at least grade 2, or grade 1 with pain).
* The participant is a pregnant or lactating woman.
* The participant has known hypersensitivity to CEP-18770, lenalidomide, thalidomide, dexamethasone, mannitol, or hydroxypropyl betadex.
* The participant received glucocorticoid therapy (prednisone >10 mg/day orally or equivalent) within the last 2 weeks prior to the first dose of study drug.
* The participant has a history of malignancy, other than multiple myeloma, within the last 5 years excluding adequately treated curable disease or indolent disease that is not likely to require therapy during the conduct of the study.
* The participant has known central nervous system (CNS) involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-08-03 (Actual); Primary Completion 2013-03-14 (Actual); Study Completion 2013-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (8):
- United States (3):
  - Teva Investigational Site 1, Augusta, Georgia
  - Teva Investigational Site 3, Lexington, Kentucky
  - Teva Investigational Site 2, Houston, Texas
- New Zealand (5):
  - Teva Investigational Site 201, Auckland
  - Teva Investigational Site 204, Auckland
  - Teva Investigational Site 200, Christchurch
  - Teva Investigational Site 206, Hamilton
  - Teva Investigational Site 205, Newtown

RESULTS

PARTICIPANT FLOW:
Groups:
- CEP-18770 Dose A: Participants received Dose A intravenously (IV) on Days 1, 8, and 15 in each 28-day cycle. In addition, participants received a fixed dose of 25 mg oral lenalidomide on Days 1 through 21 and a fixed dose of 40 mg oral dexamethasone on Days 1, 8, 15, and 22 of each 28-day cycle.
- CEP-18770 Dose B: Participants received CEP-18770 Dose B IV on Days 1, 8, and 15 in each 28-day cycle. In addition, participants received a fixed dose of 25 mg oral lenalidomide on Days 1 through 21 and a fixed dose of 40 mg oral dexamethasone on Days 1, 8, 15, and 22 of each 28-day cycle.
- CEP-18770 Dose C: Participants received CEP-18770 Dose C IV on Days 1, 8, and 15 in each 28-day cycle. In addition, participants received a fixed dose of 25 mg oral lenalidomide on Days 1 through 21 and a fixed dose of 40 mg oral dexamethasone on Days 1, 8, 15, and 22 of each 28-day cycle.
Period: Overall Study
Arm/Group | CEP-18770 Dose A | CEP-18770 Dose B | CEP-18770 Dose C
Started | 3 | 5 | 3
Received at Least 1 Dose of Study Drug | 3 | 5 | 3
Completed | 0 | 2 | 2
Not Completed | 3 | 3 | 1
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Disease progression | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set for part 1 included all participants who received at least 1 dose of CEP-18770.
Groups:
- Total: Total of all reporting groups
Arm/Group | CEP-18770 Dose A | CEP-18770 Dose B | CEP-18770 Dose C | Total
Number analyzed (Participants) | 3 | 5 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (3.06) | 61.4 (11.67) | 57.7 (15.37) | 61.2 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 4
  Male | 1 | 3 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 2 | 3 | 2 | 7
  Race: Black | 1 | 2 | 0 | 3
  Race: Asian | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) in Participants Treated at the (Maximum Tolerated Dose) MTD, as Assessed Using International Myeloma Working Group (IMWG) Criteria
Description: The ORR is defined as percentage of participants who achieve a best response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) during the study. sCR: negative immunofixation in serum and urine; disappearance of any soft tissue plasmacytomas; < 5% plasma cells in bone marrow; normal free light chain (FLC) ratio; and absence of clonal cells in bone marrow. CR: negative immunofixation in serum and urine; disappearance of any soft tissue plasmacytomas; and <5% plasma cells in bone marrow. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis; 90% or greater reduction in serum M-protein level and urine M-protein level less than 100 milligrams (mg)/24 hours. PR: ≥50% reduction in serum M-protein level; ≥90% reduction in 24-hour urinary M-protein level or reduction to less than 200 mg per 24 hours; and ≥50% reduction in the size of any soft tissue plasmacytomas present at baseline.
Time Frame: From the first administration of CEP-18770 up to approximately 1.5 years
Population: The full analysis set included all participants who received at least 1 dose of CEP-18770 at the MTD, including participants treated at the MTD of CEP-18770 in Part 1 and who had at least 1 response assessment, or who discontinued treatment due to toxicity or death. Participants who did not have a response assessment were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CEP-18770 Dose B
Number analyzed (Participants) | 5
percentage of participants | 40 [5.27 to 85.34]

2. Primary Outcome: Maximum Tolerated Dose of CEP-18770
Description: MTD was based on the assessment of dose-limiting toxicity (DLT) during cycle 1 only and was defined as the highest dose at which fewer than one-third of participants in a cohort experience DLT. A DLT was defined as any of the following drug-related toxicities occurring during Cycle 1: Hematologic adverse events (AEs) (Grade 4 hematologic AEs, Grade 3 hematologic AEs with sequelae); Grade 3 nonhematologic AEs; Neuropathy (Grade 2 neuropathy, Grade 1 neuropathy with pain, worsening grade of neuropathy or new symptoms of pain associated with neuropathy); Any other toxicity that, in the judgment of the principal investigator, was a DLT; If a participant cannot receive 75% of the planned dose for any of the 3 agents (missing >1 dose of CEP-18770, or >5 doses of lenalidomide, or >1 dose of dexamethasone [either consecutively or separately]), due to a drug-related AE, the event was considered a DLT, even if the grade of toxicity was lower than specified DLT determination as described above.
Time Frame: Cycle 1 (28 days)
Population: The MTD determination set included all participants who received at least 3 doses of the study drug during the first cycle. In addition, any participant who experienced a drug related DLT during Cycle 1 was considered evaluable regardless of the number of doses received.
Measure: Number; unit: mg/m^2
Groups:
- Overall Population: Participants received CEP-18770 Dose A, Dose B or Dose C IV on Days 1, 8, and 15 in each 28-day cycle. In addition, participants received a fixed dose of 25 mg oral lenalidomide on Days 1 through 21 and a fixed dose of 40 mg oral dexamethasone on Days 1, 8, 15, and 22 of each 28-day cycle.
Arm/Group | Overall Population
Number analyzed (Participants) | 11
mg/m^2 | 1.8

3. Secondary Outcome: Duration of Response (DOR) for Participants Treated With CEP-18770 at the MTD, as Assessed Using IMWG Criteria
Description: DOR was defined as the time interval from the date of first response (sCR, CR, VGPR, or PR) to the date of disease progression. sCR, CR, VGPR, and PR as defined in outcome measure 1. Disease progression was defined as any 1 or more of the following: Increase of 25% or more from lowest response level in any 1 or more of the following: - serum M-component (absolute increase must be ≥0.5 grams [g]/deciliter [dL]), - urine M-component (absolute increase must be ≥200 mg/24 hours), bone marrow plasma cell percentage ≥10%; definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; and development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that could be attributed solely to the plasma cell proliferation disorder.
Time Frame: From the date of first response to the date of disease progression (up to approximately 1.5 years)
Population: The full analysis set included all participants who received at least 1 dose of CEP-18770 at the MTD, including participants treated at the MTD of CEP-18770 in Part 1 and who had at least 1 response assessment, or who discontinued treatment due to toxicity or death. Participants who did not have a response assessment were considered non-responders. Overall number of participants analyzed = participants with a response of sCR, CR, VGPR, or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CEP-18770 Dose B
Number analyzed (Participants) | 2
months | NA [NA to NA] — No participants with a response had an event of disease progression or death, hence the data could not be calculated.

4. Secondary Outcome: Time to Progression (TTP) for Participants Treated With CEP-18770 at the MTD, as Assessed Using IMWG Criteria
Description: TTP was defined as the time interval from the date of first dose to the date of disease progression. Disease progression was defined as any 1 or more of the following: Increase of 25% or more from lowest response level in any 1 or more of the following: - serum M-component (absolute increase must be ≥0.5 g/dL), - urine M-component (absolute increase must be ≥200 mg/24 hours), bone marrow plasma cell percentage ≥10%; definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; and development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that could be attributed solely to the plasma cell proliferation disorder.
Time Frame: From the date of first dose of study drug to the date of disease progression (up to approximately 1.5 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CEP-18770 Dose B
Number analyzed (Participants) | 5
months | NA [10.2 to NA] — Due to small number of participants with an event, median and upper limit of 95% confidence interval (CI) could not be calculated.

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: From the first administration of CEP-18770 up to approximately 1.5 years
Population: Safety analysis set included all participants who received at least 1 dose of CEP-18770.
Measure: Count of Participants; unit: Participants
Arm/Group | CEP-18770 Dose A | CEP-18770 Dose B | CEP-18770 Dose C
Number analyzed (Participants) | 3 | 5 | 3
Participants | 3 | 5 | 3

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of CEP-18770
Time Frame: Before and immediately after end of infusion (EOI) and at approximately 2, 4, and 8 hours after the EOI on Days 1 and 15 of Cycle 1
Population: The pharmacokinetic (PK) analysis set included all participants for whom at least 1 PK parameter can be calculated. Here, number analyzed = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/ milliliter (mL)
Arm/Group | CEP-18770 Dose A | CEP-18770 Dose B | CEP-18770 Dose C
Number analyzed (Participants) | 3 | 5 | 3
nanograms (ng)/ milliliter (mL)
  Day 1 | 579.49 (118.48) | 663.00 (164.84) | 876.97 (211.99)
  Day 15: number analyzed (Participants) | 3 | 5 | 1
  Day 15 | 639.59 (242.96) | 628.07 (291.34) | 977.09

7. Secondary Outcome: Time to Reach Cmax (Tmax) of CEP-18770
Time Frame: as for outcome 6
Population: The PK analysis set included all participants for whom at least 1 PK parameter can be calculated. Here, number analyzed = participants evaluable at specified timepoint.
Measure: Median (Full Range); unit: hours
Arm/Group | CEP-18770 Dose A | CEP-18770 Dose B | CEP-18770 Dose C
Number analyzed (Participants) | 3 | 5 | 3
hours
  Day 1 | 0.07 [0.03 to 0.12] | 0.08 [0.05 to 0.18] | 0.10 [0.08 to 0.13]
  Day 15: number analyzed (Participants) | 3 | 5 | 1
  Day 15 | 0.07 [0.05 to 0.08] | 0.08 [0.05 to 0.15] | 0.08 [0.08 to 0.08]

8. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to t (AUC0-t) of CEP-18770
Time Frame: as for outcome 6
Population: PK analysis set included all participants for whom at least 1 PK parameter can be calculated. Here, number analyzed = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: ng*hours/mL
Arm/Group | CEP-18770 Dose A | CEP-18770 Dose B | CEP-18770 Dose C
Number analyzed (Participants) | 3 | 5 | 3
ng*hours/mL
  Day 1 | 673 (618) | 1371 (656) | 1527 (357)
  Day 15: number analyzed (Participants) | 3 | 5 | 1
  Day 15 | 1595 (677) | 2071 (1240) | 2266

ADVERSE EVENTS:
Time Frame: From the first administration of CEP-18770 up to approximately 1.5 years
Description: Safety analysis set included all participants who received at least 1 dose of CEP-18770.
Arm/Group | CEP-18770 Dose A | CEP-18770 Dose B | CEP-18770 Dose C
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/5 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEP-18770 Dose A (N=3) | CEP-18770 Dose B (N=5) | CEP-18770 Dose C (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEP-18770 Dose A (N=3) | CEP-18770 Dose B (N=5) | CEP-18770 Dose C (N=3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (16) | 2 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (8)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 3 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 4 (4) | 3 (3)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion site phlebitis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 1 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Neutrophil percentage decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (6)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.